CLINICAL TRIAL: NCT06834035
Title: Targeting Collagen VII Antibodies With IV IgG in Dystrophic Epidermolysis Bullosa
Acronym: IV IgG
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M. Peter Marinkovich (Other)
Collaborators: Epidermolysis Bullosa Research Partnership (Other Government)
Responsible Party: Sponsor-Investigator, M. Peter Marinkovich, Associate Professor of Dermatology, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 73958
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Epidermolysis Bullosa; Epidermolysis Bullosa Acquisita; Dystrophic Epidermolysis Bullosa; Recessive Dystrophic Epidermolysis Bullosa
Keywords: Epidermolysis Bullosa; Epidermolysis Bullosa Acquisita; Dystrophic Epidermolysis Bullosa; Recessive Dystrophic Epidermolysis Bullosa; Collagen 7; C7; Col7; EB; EBA; DEB; RDEB; Antibodies; Collagen VII; IV IgG; IgG; IVIgG; C7 Antibodies; Collagen 7 Antibodies; Collagen VII Antibodies; Vyjuvek; B-VEC
MeSH Terms: conditions — Epidermolysis Bullosa; Epidermolysis Bullosa Acquisita; Epidermolysis Bullosa Dystrophica | interventions — Immunoglobulin G

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intra-Personal Control (Experimental): There is one arm of the study. First, each participant undergoes a 3-month observational period, during which they continue application of their prescribed Vyjuvek. After 3 months, they enter the treatment period, during which they continue their Vyjuvek application and, in addition, receive the IV IgG treatment.
  Interventions: Biological: Immunoglobulin G

INTERVENTIONS:
Biological: Immunoglobulin G — Purified IgG from human serum, delivered via IV
  Other Names: IgG; IV IgG

SUMMARY:
The study objective is to see if IV IgG treatment in Recessive Dystrophic Epidermolysis Bullosa (RDEB) skin in conjunction with VYJUVEK treatment improves wound healing and affects the levels of C7 and HSV-1 antibody levels in serum.

Fewer wounds, more rapidly healing wounds, and decreased C7 and HSV-1 antibodies could improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of generalized Recessive dystrophic epidermolysis bullosa (RDEB) demonstrated by COL7A1 mutations.
2. Diagnosis of EBA demonstrated by the presence of levels of serum C7 antibodies above the normal ELISA range
3. Baseline skin blistering greater than 5% total body surface area
4. 1 wound at least 20 cm^2 able to be entirely treated with Vyjuvek weekly
5. 1 wound at least 20 cm^2 that has never been treated with Vyjuvek
6. Ongoing VYJUVEK treatment.

Exclusion Criteria:

1. History of thrombotic event(s)
2. History of cardiac failure
3. History of renal failure
4. IgA deficiency

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-08-04 (Estimated); Primary Completion 2026-03-06 (Estimated); Study Completion 2026-03-06 (Estimated)

PRIMARY OUTCOMES:
Adverse Events and Effects | 9 Months
  Occurrence of adverse events and effects
Percent Change in Wound Area | 9 Months
  The wound area at the end of the treatment phase compared to the wound area at the beginning of the treatment phase.
  Wound healing (% and cm^2) over the course of the treatment phase compared to the wound healing (% and cm^2), over the observation phase.

CONTACTS AND LOCATIONS:
Overall Officials: Matt P Marinkovich, MD, Principal Investigator — Associate Professor of Dermatology
Locations (1):
- Stanford University, Redwood City, California, United States